CLINICAL TRIAL: NCT04506073
Title: A Randomized, Double-blind, Placebo-controlled Trial of Allogeneic Bone Marrow-derived Mesenchymal Stem Cells as a Disease-modifying Therapy for Idiopathic Parkinson's Disease
Brief Title: Phase IIa Randomized Placebo Controlled Trial: Mesenchymal Stem Cells as a Disease-modifying Therapy for Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Mya Schiess, Professor and Adriana Blood Chair in Neurology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-20-0150
Record Dates: First submitted 2020-07-16; First posted 2020-08-10 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Parkinson's Disease
Keywords: Stem Cells; Mesenchymal stem cells; Inflammatory markers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mesenchymal Stem Cells and Placebo (Experimental): 2 infusions of 10 X 10^6 MSC/kg and 1 placebo infusion, all doses administered 4 months apart.
  Interventions: Drug: Mesenchymal Stem Cells; Drug: Placebo
- Mesenchymal Stem Cells (Experimental): 3 infusions of 10 X 10^6 MSC/kg administered every 4 months.
  Interventions: Drug: Mesenchymal Stem Cells
- Placebo (Placebo Comparator): 3 placebo doses administered every 4 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesenchymal Stem Cells — 1 dose is 10 X 10^6 MSC/kg
  Other Names: allogeneic mesenchymal stem cells
  Arms: Mesenchymal Stem Cells; Mesenchymal Stem Cells and Placebo
Drug: Placebo — Placebo will be identical to the investigational product but will not contain mesenchymal stem cells (MSCs).
  Arms: Mesenchymal Stem Cells and Placebo; Placebo

SUMMARY:
The purpose of this study is to select the safest and most effective number of repeat doses of allogeneic bone marrow-derived mesenchymal stem cell (MSC) infusions to slow the progression of Parkinson's disease (PD).

DETAILED DESCRIPTION:
Single site phase IIa study of allogeneic MSC in a double blind randomized control trial as disease modifying therapy for PD. The design includes three treatment arms with 45 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease by the UK brain bank criteria including the presence of 2 cardinal signs of PD plus bradykinesia.
* Mild microsomia to anosmia.
* A modified Hoehn and Yahr stage of 3 or less.
* Date of diagnosis of PD between 3 to 10 years
* Robust response to dopaminergic therapy.

Exclusion Criteria:

* Atypical, vascular, or drug-induced Parkinsonism.
* An atypical DAT scan or MRI supporting an alternative explanation for PD symptoms.
* Patient not on levodopa containing medications.
* Clinical features of psychosis or refractory hallucinations.
* A Montreal Cognitive Assessment (MoCA) score of less than 25.
* Uncontrolled seizure disorder.
* Abnormal Kidney and liver function.
* Presence of clinically refractory orthostatic hypotension at the screening or baseline visit.
* Body mass index of greater than or equal to 35.
* Cardiac disease: History of congestive heart failure, clinically significant bradycardia, presence of 2nd, or 3rd-degree atrioventricular block.
* Pulmonary disease: COPD with oxygen-requirement at rest or with ambulation; or moderate to severe asthma.
* Active malignancy or diagnosis of malignancy within 5 years prior to the start of screening
* Any current suicidal ideation or behaviors.
* Any diagnosis of autoimmune disease or immunocompromised state
* History of medium or large size vessel cerebrovascular accidents.
* History of traumatic brain injury with loss of consciousness and residual neurologic symptoms.
* Major surgery within the previous 3 months or planned in the ensuing 6 months.
* History of use of an investigational drug within 90 days prior to the screening visit.
* History of brain surgery for PD.
* Substance abuse disorder.
* Active anticoagulation treatment and/or abnormal INR.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Safest number of effective doses of MSC as measured by the Part III of the Movement Disorder Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) scale | Screening
Safest number of effective doses of MSC as measured by the Part III of the Movement Disorder Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) scale | Week 7, post infusion #1
Safest number of effective doses of MSC as measured by the Part III of the Movement Disorder Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) scale | Week 20, post infusion #2
Safest number of effective doses of MSC as measured by the Part III of the Movement Disorder Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) scale | Week 29, post-infusion #3
Safest number of effective doses of MSC as measured by the Part III of the Movement Disorder Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) scale | Week 39 follow-up
Safest number of effective doses of MSC as measured by the Part III of the Movement Disorder Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) scale | Week 52 follow-up
Safest number of effective doses of MSC as measured by the Part III of the Movement Disorder Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) scale | Week 78 follow-up

SECONDARY OUTCOMES:
Safety and tolerability as measured by serious adverse reactions. | Baseline,week 7,week 20,week 29,week 39,week 78
Safety and tolerability as measured by immunologic responses. | Baseline,week 7,week 20,week 29,week 39,week 78
  Donor specific antibodies (DSA) in serum of patients will be measured and compared to baseline to determine if there is a development of antibody response to donor HLA (human leukocyte antigen). This will determine if there is a possibility of anti-donor alloimmune response after the first or second infusion of MSC, which might lead to a subsequent antibody-mediated rejection (AMR) with the following infusion. Testing will be done at the these time points to determine if 2nd or 3rd infusions will continue.
Motor function as measured by the Timed-Up-and-Go (TUG) scale | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
  This test uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. A longer duration of time indicates a worse outcome
Global measurement of disability as measured by the change in the screening "Off" modified Hoehn and Yahr (H&Y) | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
Quality of life as measured by the modified Schwab and England activities of daily living scale (ADL) | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
Quality of life as measured by the Parkinson's Disease Questionnaire 39 (PDQ-39) | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
Quality of life as measured by the EuroQol- 5 Dimension (EQ-5D) | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
Non-motor symtoms as measured by the The University of Pennsylvania Smell Identification Test (UPSIT- 40 odor test booklet). | Baseline,week 29,week 78
Cognitive function as measured by the the change in Montreal Cognitive Assessment (MoCA) | Baseline,week 29,week 78
Behavioral changes as measured by the Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool that evaluates suicidal ideation and behavior. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent". Exclusionary criteria views 1 or more positive answers in the last month as not eligible for participation. In follow up, one positive response requires further investigation.
Behavioral changes as measured by the Geriatric Depression Scale-Short Form (GDS-SF) | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
  The Geriatric Depression Scale Short form (GDS-SF) is a 15-item screening tool that is used to identify depression in older adults. Answers indicating depression are in bold and italicized; score one point for each bold one selected. A score of 0 to 5 is normal. A score greater than 5 suggests depression and requires evaluation, whereas a score of 10 or greater would require evaluation for treatment .
Behavioral changes as measured by the Parkinson Anxiety Scale (PAS) | Baseline,week 7,week 20,week 29,week 39,week 52,week 78
Measurement of putative paracrine mechanism of MSCs using neuroimaging | Baseline,week 29,week 78
Measurement of putative paracrine mechanism of MSCs as measured by concentration of cytokines in patient blood sample. | Baseline,week 7,week 20,week 29,week 39,week 78
  Examples of these are IL-1beta, IL-6, TNF-alpha, COX-2 and PGE-2. These are measured by Magnetic Bead Panel - Multiplex Assay or ELISA, allowing for specificity in the blood.
Measurement of putative paracrine mechanism of MSCs as measured by concentration of chemokines in patient blood sample. | Baseline,week 7,week 20,week 29,week 39,week 78
  Examples of these are CCL2 (MCP-1), CCL7 (MCP-3), CCL11 (Eotaxin) CCL2 (MDC), CXCL10 (IP-10), CX3CL1 (Fractalkine). These will be measured by Magnetic Bead Panel - Multiplex Assay or ELISA, allowing for specificity in the blood.
Measurement of putative paracrine mechanism of MSCs as measured by concentration of growth factors | Baseline,week 7,week 20,week 29,week 39,week 78
  Examples of these are Glial Derived Neurotrophic Factor, Brain Derived Neurotrophic Factor and Vascular Epidermal Growth Factor . These will be measured by ELISA specific to blood and CSF.
Measurement of putative paracrine mechanism of MSCs as measured by concentration of neurotransmitters | Baseline,week 7,week 20,week 29,week 39,week 78
  Examples of these are homovanillic acid and 5-hydroxytryptamine. These will be measured in CSF and blood by ELISA.
Measurement of putative paracrine mechanism of MSCs as measured by alpha-synuclein oligomers in the blood (serum or plasma) | Basleline,week 29,week 39,week 78
Measurement of putative paracrine mechanism of MSCs as measured by alpha-synuclein oligomers in the cerebral spinal fluid | Baseline,week 39

CONTACTS AND LOCATIONS:
Overall Officials: Mya C Schiess, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Background] Connolly BS, Lang AE. Pharmacological treatment of Parkinson disease: a review. JAMA. 2014 Apr 23-30;311(16):1670-83. doi: 10.1001/jama.2014.3654. PMID 24756517
- [Background] Jellinger KA. Basic mechanisms of neurodegeneration: a critical update. J Cell Mol Med. 2010 Mar;14(3):457-87. doi: 10.1111/j.1582-4934.2010.01010.x. Epub 2010 Jan 11. PMID 20070435
- [Background] Kortekaas R, Leenders KL, van Oostrom JC, Vaalburg W, Bart J, Willemsen AT, Hendrikse NH. Blood-brain barrier dysfunction in parkinsonian midbrain in vivo. Ann Neurol. 2005 Feb;57(2):176-9. doi: 10.1002/ana.20369. PMID 15668963
- [Background] Gray MT, Woulfe JM. Striatal blood-brain barrier permeability in Parkinson's disease. J Cereb Blood Flow Metab. 2015 May;35(5):747-50. doi: 10.1038/jcbfm.2015.32. Epub 2015 Mar 11. PMID 25757748
- [Background] Orr CF, Rowe DB, Halliday GM. An inflammatory review of Parkinson's disease. Prog Neurobiol. 2002 Dec;68(5):325-40. doi: 10.1016/s0301-0082(02)00127-2. PMID 12531233
- [Background] Nagatsu T, Mogi M, Ichinose H, Togari A. Cytokines in Parkinson's disease. J Neural Transm Suppl. 2000;(58):143-51. PMID 11128604
- [Background] Stypula G, Kunert-Radek J, Stepien H, Zylinska K, Pawlikowski M. Evaluation of interleukins, ACTH, cortisol and prolactin concentrations in the blood of patients with parkinson's disease. Neuroimmunomodulation. 1996 Mar-Jun;3(2-3):131-4. doi: 10.1159/000097237. PMID 8945728
- [Background] Joyce N, Annett G, Wirthlin L, Olson S, Bauer G, Nolta JA. Mesenchymal stem cells for the treatment of neurodegenerative disease. Regen Med. 2010 Nov;5(6):933-46. doi: 10.2217/rme.10.72. PMID 21082892
- [Derived] Martinez-Lemus JD, Molony DA, Suescun J, Tharp E, Thomas TS, Green C, Onuigbo C, Ritter R 3rd, Schiess MC. Allogeneic bone marrow-derived mesenchymal stem cells in the aging kidney: secondary results of a Parkinson's disease clinical trial. Stem Cell Res Ther. 2025 Sep 24;16(1):493. doi: 10.1186/s13287-025-04577-y. PMID 40993774